CLINICAL TRIAL: NCT03769454
Title: A Phase I Safety and Tolerability Study of PP-001 Eye Drops in Healthy Adult Volunteers
Brief Title: A Phase I Study of PP-001 Eye Drops in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Panoptes Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PP-001-1101
Record Dates: First submitted 2018-12-06; First posted 2018-12-07 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Keratoconjunctivitis; Ocular Surface Disease
MeSH Terms: conditions — Keratoconjunctivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- PP-001 verum - cohort 1 (Experimental): PP-001 verum - cohort 1
  Interventions: Drug: PP-001
- Placebo - cohort 1 (Placebo Comparator): Placebo - cohort 1
  Interventions: Other: Placebo
- PP-001 verum - cohort 2 (Experimental): PP-001 verum - cohort 2
  Interventions: Drug: PP-001
- Placebo - cohort 2 (Placebo Comparator): Placebo - cohort 2
  Interventions: Other: Placebo
- PP-001 verum - cohort 3 (Experimental): PP-001 verum - cohort 3
  Interventions: Drug: PP-001
- Placebo - cohort 3 (Placebo Comparator): Placebo - cohort 3
  Interventions: Other: Placebo
- PP-001 verum - cohort 4 (Experimental): PP-001 verum - cohort 4
  Interventions: Drug: PP-001
- Placebo - cohort 4 (Placebo Comparator): Placebo - cohort 4
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PP-001 — PP-001 eye drops
  Arms: PP-001 verum - cohort 1; PP-001 verum - cohort 2; PP-001 verum - cohort 3; PP-001 verum - cohort 4
Other: Placebo — Placebo eye drops
  Arms: Placebo - cohort 1; Placebo - cohort 2; Placebo - cohort 3; Placebo - cohort 4

SUMMARY:
In this study, PP-001 eye drops are assessed for safety and tolerability in healthy, adult volunteers. PP-001 is a novel, anti-inflammatory small molecule that inhibits a specific enzyme (Dihydroorotate Dehydrogenase).

The study was amended and now includes patients with ocular surface inflammation.

DETAILED DESCRIPTION:
In this prospective, single-centre, double blind (within each cohort), placebo controlled, randomised study, safety and tolerability of PP-001 eye drops is assessed in healthy, adult volunteers (cohorts 1-3) and in patients with ocular surface inflammation (cohort 4). PP-001 is a novel small molecule inhibitor of Dihydroorotate Dehydrogenase (DHODH) with anti-inflammatory properties.

ELIGIBILITY:
Inclusion Criteria (excerpt):

Cohorts 1-3:

* male or female healthy volunteers 18 - 64 years of age
* good general state of health and participants must not have a diagnosis of any eye disease that could effect the pharmacokinetics of PP-001

Cohort 4:

* male or female subjects 18-64 years of age with ocular surface inflammation in both eyes
* ocular surface inflammation as defined per protocol
* good general state of health

Exclusion Criteria (excerpt):

Cohorts 1-4:

* participation in other clinical trials within 30 days prior to dosing start (ocular and non-ocular clinical trials)
* pregnant or nursing patients
* regular use of any ocular agents within 60 days prior to start dosing

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety and tolerability by determining treatment emergent adverse events | 28 days (cohorts 1-3) and 20 days (cohort 4)
  To assess safety and tolerability of ascending, multiple daily doses of PP-001 eye drops in healthy, adult volunteers and in patients with ocular surface inflammation

SECONDARY OUTCOMES:
Evaluation of Peak Plasma Concentration (Cmax) in peripheral blood | 1 and 12 days (cohorts 1-3)
  To evaluate the pharmacokinetics (Cmax) of PP-001 in healthy, adult volunteers following single and multiple daily ocular instillation
Evaluation of area under the plasma concentration versus time curve (AUC) in peripheral blood | 1 and 12 days (cohorts 1-3)
  To evaluate the pharmacokinetics (AUC) of PP-001 in healthy, adult volunteers following single and multiple daily ocular instillation

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Vienna, Vienna, Austria

DOCUMENTS (2):
  • Study Protocol (2021-03-26): https://cdn.clinicaltrials.gov/large-docs/54/NCT03769454/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/54/NCT03769454/SAP_001.pdf